CLINICAL TRIAL: NCT01684410
Title: A Three Week Dose Escalation, Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Safety and Tolerability of 100 mg or 200 mg of Inhaled Alpha-1 HC, Once a Day in Subjects With Cystic Fibrosis.
Brief Title: Safety and Tolerability Trial of Inhaled Alpha1-Proteinase Inhibitor (Human), Hydrophobic Chromatography Process (Alpha-1 HC) in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T6005-201
Record Dates: First submitted 2012-09-06; First posted 2012-09-13 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Alpha1-proteinase inhibitor; Alpha1-antitrypsin
MeSH Terms: conditions — Cystic Fibrosis; alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alpha-1 HC 100 mg (Experimental): 100 mg of aerosolized Alpha-1 HC inhaled daily via nebulizer for 3 weeks.
  Interventions: Biological: Alpha-1 HC 100 mg
- Alpha-1 HC 200 mg (Experimental): 200 mg of aerosolized Alpha-1 HC inhaled daily via nebulizer for 3 weeks.
  Interventions: Biological: Alpha-1 HC 200 mg
- Placebo (Placebo Comparator): Placebo inhaled daily via nebulizer for 3 weeks. Placebo (phosphate buffer saline with polysorbate).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Alpha-1 HC 100 mg — Alpha-1 HC is a sterile, liquid preparation of purified alpha1-proteinase inhibitor prepared from pooled human plasma. Alpha-1 HC 100 mg inhaled once daily for 21 days for a total of 21 inhaled treatments.
  Other Names: Alpha1-proteinase inhibitor; alpha1-antitrypsin
  Arms: Alpha-1 HC 100 mg
Biological: Placebo — Phosphate Buffer Saline with Polysorbate (placebo) composed of the same elements listed for Alpha-1 HC, minus the 50 mg/mL of Alpha-1 HC. Placebo inhaled once daily for 21 days for a total of 21 inhaled treatments.
  Arms: Placebo
Biological: Alpha-1 HC 200 mg — Alpha-1 HC is a sterile, liquid preparation of purified alpha1-proteinase inhibitor prepared from pooled human plasma. Alpha-1 HC 200 mg inhaled once daily for 21 days for a total of 21 inhaled treatments.
  Other Names: Alpha1-proteinase inhibitor; alpha1-antitrypsin
  Arms: Alpha-1 HC 200 mg

SUMMARY:
This was a randomized, double-blind, placebo-controlled, dose escalation study to assess the safety and tolerability of 100 mg and 200 mg of inhaled Alpha-1 HC administered once a day for three weeks in subjects aged 18 years and older with cystic fibrosis (CF). The treatment duration in this study was intended to provide multi-dose safety information prior to proceeding to longer durations of exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Documentation of CF diagnosis.
* Have a pre-bronchodilator FEV1 ≥ 40% of predicted at Visit 1 and have a Visit 2 pre-investigational product FEV1 that is ≥ 40% of predicted and within ± 15% of the Visit 1 result.
* Deemed by the Investigator to be a suitable candidate for serial collection of expectorated sputum.

Exclusion Criteria:

* Had a pulmonary exacerbation during the 4 weeks before screening (Visit 1) which required the initiation of new antibiotic treatment
* Have a pulmonary exacerbation during the screening period (between Visit 1 and Visit 2) which requires the initiation of new antibiotic treatment
* FEV1 < 0.59 liters at the screening visit
* Respiratory insufficiency with continuous supplemental oxygen therapy, or carbon dioxide retention
* Elevated aspartate transaminase (AST) or alanine aminotransferase (ALT) that is ≥ 3 times the upper limit of normal for age and gender
* Smoking during the past 6 months
* Lung surgery during the past 2 years
* Positive culture for Burkholderia cepacia or mycobacterium during the past two years.
* Active allergic bronchopulmonary aspergillosis
* Pre-treatment sputum collection at Visit 1 or Visit 2 (Randomization) characterized by problems such as inadequate sputum volume or quality.
* Known selective Immunoglobulin A (IgA) deficiency with known antibody against IgA (anti-IgA antibody).
* History of anaphylaxis or severe systemic response to any plasma-derived alpha1-proteinase inhibitor preparation or other blood product(s), or to polysorbates.
* Use of chronic oral steroids during the study. Note: Inhaled corticosteroids that had been administered for at least 4 weeks prior to Visit 1 were permissible during the study.
* Use of chronic, high dose ibuprofen therapy within 3 weeks of screening and at anytime during the study.
* Chronic maintenance therapy with systemic antibiotics within 3 weeks of screening and through last dose of investigational product.
* Use of leukotriene synthesis inhibitor (zileuton) or leukotriene receptor antagonists (montelukast, zafirlukast) within 3 weeks of screening and at anytime during the study.
* Use of roflumilast within 3 weeks of screening and at any time during the study.
* Initiation of a new chronic medication or dosage change of a chronic medication for treatment of cystic fibrosis (example: Kalydeco™ [ivacaftor]) within 3 weeks of screening (Visit 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - National Jewish Hospital, Denver, Colorado
  - Children's Hospital Boston, Boston, Massachusetts
  - UNC at Chapel Hill, Chapel Hill, North Carolina
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 41 subjects provided informed consent and were screened for the study. Eleven (11) subjects were screen failures, and a total of 30 subjects were randomized to one of three treatment groups: 200 mg or 100 mg of Alpha-1 HC or placebo daily.
Groups:
- Alpha-1 HC 100 mg: 100 mg of aerosolized Alpha-1 HC inhaled daily via nebulizer for 3 weeks.
  Alpha-1 HC: Alpha-1 HC is a sterile, liquid preparation of purified alpha1-proteinase inhibitor prepared from pooled human plasma.
- Alpha-1 HC 200 mg: 200 mg of aerosolized Alpha-1 HC inhaled daily via nebulizer for 3 weeks.
  Alpha-1 HC: Alpha-1 HC is a sterile, liquid preparation of purified alpha1-proteinase inhibitor prepared from pooled human plasma.
- Placebo: Placebo inhaled daily via nebulizer for 3 weeks. Placebo (phosphate buffer saline with polysorbate).
  Placebo
Period: Overall Study
Arm/Group | Alpha-1 HC 100 mg | Alpha-1 HC 200 mg | Placebo
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) Population: included all subjects who were randomized (included those withdrawn from treatment for any reason).
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpha-1 HC 100 mg | Alpha-1 HC 200 mg | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (10.62) | 28.1 (11.43) | 29.3 (9.96) | 28.5 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 6 | 20
  Male | 2 | 4 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: adverse event frequency
Time Frame: 3 weeks
Population: Safety Population: included all subjects who received any dose of IP (included those withdrawn from treatment for any reason)
Measure: Number; unit: percentage of participants
Arm/Group | Alpha-1 HC 100 mg | Alpha-1 HC 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
percentage of participants | 100 | 80 | 60

2. Other Pre Specified Outcome: Percent Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 3
Description: FEV1 conducted before and after inhalation of the investigational product at study visits.
Time Frame: 3 weeks
Population: Safety Population: included all subjects who received any dose of Investigational Product (included those withdrawn from treatment for any reason)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Alpha-1 HC 100 mg | Alpha-1 HC 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
percent | 1.5 (5.20) | -2.1 (12.28) | 0.5 (5.91)

3. Other Pre Specified Outcome: Percent Change From Baseline in Forced Vital Capacity (FVC) at Week 3
Description: FVC conducted before and after inhalation of the investigational product
Time Frame: 3 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Alpha-1 HC 100 mg | Alpha-1 HC 200 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
percent | 1.2 (5.23) | -2.3 (11.57) | -0.9 (3.73)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Alpha-1 HC 100 mg | Alpha-1 HC 200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 10/10 | 8/10 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-1 HC 100 mg (N=10) | Alpha-1 HC 200 mg (N=10) | Placebo (N=10)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EXACERBATION/ (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-1 HC 100 mg (N=10) | Alpha-1 HC 200 mg (N=10) | Placebo (N=10)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 2 (2) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 1 (1)
ORAL HERPES (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BREATH SOUNDS ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
FORCED EXPIRATORY VOLUME DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
PHYSICAL EXAMINATION ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0)
PULMONARY FUNCTION TEST DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
SPUTUM ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SINUS HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
BRONCHIAL SECRETION RETENTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
PHARYNGEAL ERYTHEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PHARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
PULMONARY EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
RALES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
RESPIRATORY TRACT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RHONCHI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 2 (2)
OTITIS EXTERNA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.